CLINICAL TRIAL: NCT05599750
Title: A Modern Comparison of Suture Repair With Mesh Repair for Incisional Hernia
Brief Title: Suture Repair vs Mesh Repair for Incisional Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clayton Petro (Other)
Responsible Party: Sponsor-Investigator, Clayton Petro, Assistant Professor, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-945
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to intervention. Recurrence on imaging will be assessed by blinded assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hernia repair with mesh (Control arm) (Active Comparator): Participants will undergo incisional hernia repair with prolene mesh in the retrorectus position with at least 4cm of overlap.
  Interventions: Procedure: Incisional hernia repair
- Primary closure (Intervention arm) (Active Comparator): Participants will undergo incisional hernia repair with suture alone using modern surgical techniques.
  Interventions: Procedure: Incisional hernia repair

INTERVENTIONS:
Procedure: Incisional hernia repair — Participants will undergo incisional hernia repair

SUMMARY:
The goal of this randomized controlled trial is to compare the difference in quality of life at one year postoperatively for patients undergoing incisional hernia repair with mesh versus suture repair using modern techniques.

The main question it aims to answer are:

• Determine if primary suture repair is non-inferior to mesh repair for incisional hernias 2-6cm with respect to quality of life using the HerQLes summary score at one year postoperatively.

DETAILED DESCRIPTION:
This is a patient-blinded randomized control trial comparing incisional hernia repair using synthetic mesh versus suture repair. This is a non-inferiority trial theorizing that suture repair will be non-inferior with respect to quality of life (using the HerQLes survey) at 1 year postoperatively. Patients will be blinded to the intervention, groups will be in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old.
* Anticipated hernia defect 2-6cm in width
* Non-emergent case
* CDC class I
* Patients who previously underwent primary ventral hernia repair without the use of mesh
* Incisional hernia

Exclusion Criteria:

* Emergent cases
* Patients < 18 years old
* Patients who are pregnant
* Patients who previously underwent a prior ventral hernia repair with mesh at the site of the intended repair. Abdominal mesh in separate locations would be allowed.
* Ventral hernia <2cm or > 6 cm in width
* Primary hernia
* CDC wound class II-IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Hernia specific quality of life | 1 year
  Suture repair will be compared to mesh repair for incisional hernias 2-6cm with respect to quality of life using the Hernia-specific Quality of Life (HerQLes) summary score at one year postoperatively. This is reported as a score from 0-100 with higher numbers indicating better quality of life.

SECONDARY OUTCOMES:
Hernia specific quality of life | 5 years
  Compare HerQLes summary score at baseline, 30-day, and 2-year follow-up, and 5-year follow up
PROMIS-3a-Pain Intensity scores | 5 years
  Compare PROMIS-3a-Pain Intensity scores (a validated measure of pain) at baseline, 30-day, 1-year, 2 years, and 5- year follow up. Scores are reported as raw values from 3-15 or as T-scores from 30.7-71.8, with higher numbers indicating more pain.
Recurrence | 5 years
  Compare composite recurrence using clinical, radiographic exam, and Hernia Recurrence Inventory (HRI) at 1-year, and 2-year, and 5 year follow-up postoperatively
Complications | 5 years
  Compare all complications at 30-day, 1-year, 2-year, and 5-year follow-up postoperatively. This includes occurrence of surgical site infections, surgical site occurrence requiring intervention, readmissions, hernia related reoperation, or mortality.
Overall quality of life | 5 years
  4. Compare Euro-QOL-5D-5L with VAS assessment scores at baseline, 30-day, 1-year, 2 years, and 5-year follow-up.
Cost effectiveness | 5 years
  5. Perform a formal cost effectiveness analysis utilizing quality adjusted life years and incremental cost effectiveness ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Petro, MD, Principal Investigator — The Cleveland Clinic
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Northwestern, Chicago, Illinois
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Maskal SM, Miller BT, Ellis RC, Beffa LRA, Prabhu AS, Rosen MJ, Krpata DM, Huang LC, Petro CC. A modern comparison of suture repair versus mesh repair for incisional hernia: a study protocol for a randomized controlled trial. Trials. 2025 Oct 29;26(1):450. doi: 10.1186/s13063-025-08924-5. PMID 41163187